CLINICAL TRIAL: NCT02641275
Title: Self-management Training for Parents With Chronic Muscular Dystrophia
Acronym: ZRM-CMD-P
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We could not enrole or recruite enough participants.
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ZRM-CMD Parents
Record Dates: First submitted 2015-11-09; First posted 2015-12-29 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Muscular Dystrophies
Keywords: Parental stress; Muscular Dystrophies; Coping; Parental support
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Structured self-management-training (incl. systemic analysis, coaching, teaching) in 4 sessions.
  Interventions: Other: Structured self-management-training
- Control group (No Intervention): no intervention other than existing support (see exclusion criteria). However, intervention will be offered and studied secondary as well (after 1 1/2 year of no intervention).

INTERVENTIONS:
Other: Structured self-management-training — Structured self-management-training (incl. systemic analysis, coaching, teaching) in 4 sessions
  Arms: Intervention

SUMMARY:
The relentless progressive process of muscular dystrophy requires extraordinary medical, physical, and emotional care with severe consequences for caring parents (increased stress and diminished social, psychological and physical well-being). Despite the obvious need of support for parents only few and weak data exist regarding efficiency and efficacy of specific interventions supporting parental resilience and coping strategies. The presenting study aims to fill this gap by evaluating the efficacy of a structured self-management training for parents of children with severe progressive muscular dystrophy compared to parents receiving treatment as usual (TAU). In addition, investigators measure established biomarkers of psychosocial stress, such as pro-inflammatory cytokines, which will be used to monitor physiological changes with assumed significance for parental health.

DETAILED DESCRIPTION:
Background:

The relentless progressive process of muscular dystrophy requires extraordinary medical, physical, and emotional care. As a consequences caring for a patient with a severe chronic illness has been associated with increased stress and diminished social, psychological and physical well-being in parents. According to Thompson et al. 57% of parents with Duchenne muscular dystrophy children have self-reported poor psychological adjustment and, even in comparison with parents of children with other burdens like cerebral palsy or renal diseases, muscular dystrophy was associated with a wider spectrum of problems and parental stress. Moreover, parents are shown to have significant stress by feelings of guilt and associated difficulty discussing death issues with their children.

However, despite the obvious need of support for parents only few and weak data exist regarding efficiency and efficacy of specific interventions supporting parental resilience and coping strategies. In practice, they are mostly limited to meetings of self-help groups and casual exchange between concerned parents, which is rather a problem-centered than proactive solution-focused approach. As a consequence, investigators see a great need for studies regarding more specific interventions supporting parents' self-management skills, coping strategies and competencies.

Objectives:

The present study evaluates the efficacy of a structured self-management training for parents of children with severe progressive muscular dystrophy compared to parents receiving treatment as usual (TAU). In addition, investigators measure established biomarkers of psychosocial stress, such as pro-inflammatory cytokines, which will be used to monitor physiological changes with assumed significance for parental health.

Methods:

Participants will fill out online-questionnaires before, during and after self-management training. Training interventions will take place in Zurich as group sessions (10-20 participants per group). Investigators aim for a total of 60-80 participants. Parent-couples or single participants will be randomized in an intervention group (participants receiving self-management training) and a non-intervention group (participants continue with already established support). After one year parents from the non-intervention group will change into the intervention group with self- management training as well. Questionnaires focus on assessing parental strain and self- efficacy and will take 30-45minutes for each of four surveys. Validated biological markers such as cumulative cortisol levels in hair and pro-inflammatory cytokines in the blood will be collected before and after self-management trainings.

ELIGIBILITY:
Inclusion Criteria:

* Parents with at least one living child affected by chronic muscular dystrophy

Exclusion Criteria:

* Dying of a child during intervention and analysis.
* Severe/significant psychological disorder (in case of existing psychological support, participation should be agreed/supported by therapist, too)
* Recent or concomitant self-management training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Action Orientation Questionnaire (HAKEMP) | 1 1/2 year with control group
  Kuhl and co-workers introduced a special questionnaire (HAKEMP) to assess the tendency of people in concrete situations to revert to an action-oriented or state-oriented condition in 24 items.
Self-efficacy: Thought control of action (SWE) | 1 1/2 year with control group
  Quantify improved parental resilience and coping strategies facing chronic stress. Questionnaire developed by Jerusalem and Schwarzer, 1981, revised 1999 to test general self-efficacy in 10 items.
Change in Experiencing and Behaviour post-intervention (VEV) | 1 1/2 year with control group
  VEV is a questionnaire developed by Ziele and Kopf-Mehnert, 1978 to test post-intervention change in experiencing and behavior along with a retrospective life-event checklist and a self-rating questionnaire in 42 items. Other than previous questionnaires VEV will be applied only after intervention.

SECONDARY OUTCOMES:
Number of Participants With Sum of Abnormal Laboratory Values Concerning Biomarkers of psychosocial stress | 1 1/2 year with control group
  Significant lower levels of biomarkers of psychosocial stress, i.e. pro-inflammatory cytokines, which can be used to monitor physiological changes with assumed significance for parental health: C-reactive Protein (hsCRP), Tumor-Necrose-Factor alpha (TNFα), Interleukin (IL)-1ß, IL-6, und Interferon Gamma (IFNγ). Items will be aggregated as a numerical factor which shows the difference of a measured value from a reference value . Abnormal laboratory values therefore will be used as a sum.

CONTACTS AND LOCATIONS:
Overall Officials: Jürg C Streuli, MD PhD, Principal Investigator — University Children's Hospital, Zurich